CLINICAL TRIAL: NCT00515645
Title: Cardiac Autonomic Functions During Head-out Immersion and During Head Down Tilt
Acronym: IMMERSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0708061; 2007-A00727-46 (Other: AFSSAPS)
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Autonomic nervous system; Immersion; Heart rate variability; Head-down tilt; Healthy volunteers
MeSH Terms: interventions — Head-Down Tilt; Immersion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Head-down tilt and immersion

INTERVENTIONS:
Other: Head-down tilt and immersion — Head-down tilt -6° at inclusion, head-down tilt -15° at week one and Water Immersion at week two

SUMMARY:
Head down tilt (HDT) was widely used to simulate microgravity effects on cardiovascular system. HDT could be a suitable model of water immersion (WI) which is also used to simulate the cardiovascular effects of microgravity and which is not easy to study in laboratory. To define the possibility to simulate immersion by HDT, a comparison between these models is required. A comparison between WI and few angles during HDT seems necessary to understand which angle is more adapt.

The immersion induces an increase of the central blood volume. This increase is caused by a redistribution of blood from peripheral portions of the body to the intrathoracic circulation. It seems to load cardiopulmonary and arterial baroreceptors. These baroreceptors bring into play autonomic nervous system (ANS) activation and induce a bradycardia.

HDT induces an increase in central blood volume as supported by the central venous pressure and cardiac volume increase and in return, MSNA and heart rate decrease. These cardiovascular effects seem to be the same as the thermoneutral immersion and suggest that the ANS activation is the same during HDT and WI.

Nevertheless, a few previous studies about ANS in HDT indicate some discordant results: a sympathetic decrease was reported but several results show an increase of parasympathetic activity linked with a trend of increase of arterial baroreflex. The aim of this study is to assess ANS activity in HDT on different angles (-6° and -15°) and WI. The investigators suppose an increase of parasympathetic activity during WI corresponding to parasympathetic activation during HDT especially at -6°.

ELIGIBILITY:
Inclusion Criteria:

* Sportsman
* None coffee, alcohol, cigarettes 6 hours before the start of each visit
* Each meal must have been taken 4 hours before each visit
* No intensive sport 48 hours before ech visit
* Written inform consent

Exclusion Criteria:

* Subject with cardiovascular,renal disease or with metabolic syndrome
* Subject with medication
* Subject who participated to an other medical research

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
heart rate variability | inclusion, one week, two weeks

SECONDARY OUTCOMES:
Blood pressure variability | inclusion, one week, two weeks
Spontaneous baroreflex activity | inclusion, one week, two weeks
Pulmonary diffusion | inclusion, one week, two weeks
Upper limbs vascular resistance | inclusion, one week, two weeks
post ischemic forearm hyperemia | inclusion, one week, two weeks
Hematocrit rate | Inclusion, one week, two weeks
Cardiac haemodynamic | Inclusion, one week, two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Roche, MD PhD, Principal Investigator — Centre Hospitalier de Saint-Etienne
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Background] Gabrielsen A, Johansen LB, Norsk P. Central cardiovascular pressures during graded water immersion in humans. J Appl Physiol (1985). 1993 Aug;75(2):581-5. doi: 10.1152/jappl.1993.75.2.581. PMID 8226455
- [Background] Shiraishi M, Schou M, Gybel M, Christensen NJ, Norsk P. Comparison of acute cardiovascular responses to water immersion and head-down tilt in humans. J Appl Physiol (1985). 2002 Jan;92(1):264-8. doi: 10.1152/jappl.2002.92.1.264. PMID 11744669
- [Background] Ueno LM, Miyachi M, Matsui T, Takahashi K, Yamazaki K, Hayashi K, Onodera S, Moritani T. Effect of aging on carotid artery stiffness and baroreflex sensitivity during head-out water immersion in man. Braz J Med Biol Res. 2005 Apr;38(4):629-37. doi: 10.1590/s0100-879x2005000400018. Epub 2005 Apr 13. PMID 15962190